CLINICAL TRIAL: NCT05140577
Title: Reliability and Validity of the Measurement Procedure for the Evaluation of Hip Abductors Strength in Unipodal Standing Position
Brief Title: Reliability and Validity of the Evaluation of Hip Abductors Strength (RAVEHABDS)
Acronym: RAVEHABDS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: HES-SO Valais-Wallis (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01829
Record Dates: First submitted 2021-11-22; First posted 2021-12-01 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy People
Keywords: hip abductors strengthening; one-leg standing; maximal voluntary isometric strengthening; rate of force generated; dynamometer; aged category; so surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 18-30 years old: Subjects in this group is aged between 18 ans 30 years old
  Interventions: Other: Maximal voluntary isometric strengthening
- 31-65 years old: Subjects in this group is aged between 31 ans 65 years old
  Interventions: Other: Maximal voluntary isometric strengthening
- 65+ years old: Subjects in this group is aged over 65 years old
  Interventions: Other: Maximal voluntary isometric strengthening

INTERVENTIONS:
Other: Maximal voluntary isometric strengthening — The subject is asked to perform a maximum voluntary isometric force work against a wall during 5 seconds

SUMMARY:
The aim is to evaluate the intra- and inter-tester reliability, construct validity and feasibility of a new functional measurement procedure in a closed chain position on one leg. For this purpose, we will test the maximal voluntary isometric force, as well as the muscular contraction speed of the hip abductor muscles.

DETAILED DESCRIPTION:
Within this Master thesis project, we will investigate intra- and inter-tester reliability, as well as construct validity of a measurement procedure to assess hip abductor strength in a closed-chain position. Additionally, we aim to investigate some aspects of feasibility using a questionnaire about the measurement procedure and by evaluating if the test can be completing in a suitable timeframe for practical use.

To investigate intra- and inter-tester reliability, as well as construct validity, we will analyze and compare the maximal voluntary isometric strength (MVIS) and the rate of force generated (RFG) of the three groups of healthy participant (group 1: 18-30 years old; group 2: 31-65 years old; group 3: 65+ years old).

ELIGIBILITY:
Inclusion Criteria:

* Persons over 18 years old, good understanding of French, German, English or Italian, with the capacity of discernment regarding their own participation in the study

Exclusion Criteria:

* Persons with cognitive impairment or who are unable to take their own decisions about participation in the study, or who have undergone surgery on the lower limb or lumbopelvic area during the last 6 months that could contradict or influence the strength tests, will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects will be healthy adults belonging to the three age groups mentioned above
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-06-05 (Estimated)

PRIMARY OUTCOMES:
Intra-tester Correlation | 1 March, 2022
  Strength of correlation the measured values
Inter-tester correlation | 1 March, 2022
  Strength of correlation the measured values
Construct validity | 1 March, 2022
  Difference between groups by comparing values

SECONDARY OUTCOMES:
Feasibility of the measurement procedure | 1 March, 2022
  Through the administration of a feasibility questionnaire we investigate the time to perform the test, the understanding of the instructions, the fatigue, the possible pain, or the fear of falling during the test

CONTACTS AND LOCATIONS:
Locations (1):
- Sport Medical Center Ittigen, Ittigen, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of our data will be done on request